CLINICAL TRIAL: NCT03527251
Title: A Phase I Study Evaluating the Safety and Efficacy of CTLA-4 Antibody Ipilimumab Followed by PD-1 Antibody SHR-1210 in Patients With Recurrent or Metastatic Non-small Cell Lung Cancer
Brief Title: Anti-CTLA-4 Antibody Followed by Anti-PD-1 Antibody in Recurrent or Metastatic NSCLC
Acronym: SEQUENCE
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li Zhang, MD, Director of Department of Medical Oncology, Professor, Sun Yat-sen University
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2018-FXY-032
Record Dates: First submitted 2018-04-28; First posted 2018-05-17 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Non Small Cell Lung Cancer
Keywords: clinical trial, phase I; CTLA-4 antibody; PD-1 antibody; non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Ipilimumab; camrelizumab

STUDY DESIGN:
Intervention Model Description: Patients received two doses of intravenous ipilimumab (at a dose of 1 mg per kilogram of body weight) every 3 weeks, following by intravenous SHR-1210 (at a fixed dose of 200mg) every 2 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Sequential group (Experimental): intravenous ipilimumab following by intravenous SHR-1210
  Interventions: Drug: Ipilimumab; Drug: SHR-1210

INTERVENTIONS:
Drug: Ipilimumab — Patients received two doses of intravenous ipilimumab (at a dose of 1 mg per kilogram of body weight) every 3 weeks, following by intravenous SHR-1210 (at a fixed dose of 200mg) every 2 weeks.
  Other Names: Yervoy
Drug: SHR-1210 — Patients received two doses of intravenous ipilimumab (at a dose of 1 mg per kilogram of body weight) every 3 weeks, following by intravenous SHR-1210 (at a fixed dose of 200mg) every 2 weeks.

SUMMARY:
Immunotherapy has made rapid progress in melanoma, Hodgkin's lymphoma, non-small cell lung cancer, and bladder cancer, etc. Preclinical data suggested that the use of anti-PD-1 antibody in combination with CTLA-4 receptor blockers may increase antitumor activity. The CheckMate-012 study showed that nivolumab and ipilimumab combination therapy achieved an overall response rate of 43% in unselected patients with non-small cell lung cancer, compared with 23% in the nivolumab monotherapy group; and in the PD-L1 positive subgroup, nivolumab in combination with ipilimumab showed a response rate of 57%, while nivolumab alone was 28%. This showed that the combination therapy of nivolumab and ipilimumab can increase the efficacy, but the adverse events of grade 3 or above of combination therapy reach 37%. The toxic side effects limit the widespread use of nivolumab in combination with ipilimumab therapy.

However, since the action of ipilimumab is limited to the initiation of the immune response (antigen presentation and immune cell activation), and its long half-time of 15.4 days, ipilimumab can used as an induction therapy, following by the PD1 monoclonal antibody. This phase I study is aimed to evaluated the safety and efficacy of CTLA-4 antibody followed by PD-1 antibody in patients with recurrent or metastatic non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years old, male or female;
* Histologically confirmed locally advanced or metastatic non-small-cell lung cancer;
* At least one systemic chemotherapy regimen for locally advanced or metastatic disease (patients received neoadjuvant chemotherapy, concurrent chemoradiotherapy, or adjuvant chemotherapy within 6 months can be considered as first-line system therapy);
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1;
* At least one measurable lesion according to criteria RECIST v1.1;
* Life expectancy of at least 12 weeks;
* Patient has adequate bone marrow as defined by the following laboratory values:

White blood cell ≥ 3.0 × 109/L Absolute neutrophil count ≥ 1.5 × 109/L Platelets ≥ 75 × 109/L

* Patient has adequate organ function as defined by the following laboratory values:

In absence of liver metastases, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) should be below 2.5 × ULN. If the patient has liver metastases, ALT and AST should be < 5 × ULN Total serum bilirubin < ULN; or total bilirubin ≤ 3.0 × ULN with direct bilirubin within normal range of the central laboratory in patients with well documented Gilbert's Syndrome Serum creatinine ≤ 1.5 × ULN

* Provide written, informed consent to participate in the study and follow the study procedures;
* Women of childbearing potential must agree and commit to the use of a highly effective non-hormonal method of contraception, ie, intrauterine device, bilateral tubal ligation, vasectomized partner, or abstinence (only when it is the preferred lifestyle of the patient), from the time of informed consent until 28 days after the last dose of the investigational products. Men and their female partners of childbearing potential must agree and commit to use a highly effective method of contraception (ie, any of the above methods or hormonal contraception associated with inhibition of ovulation) while on treatment and for 3 months after last dose of investigational products

Exclusion Criteria:

* Driver gene EGFR, ALK and ROS were positive;
* In presence of active autoimmune disease or a history of autoimmune disease (such as the following, but not limited to: interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism, hypothyroidism; Patients with hormone replacement therapy can be included; Patients with vitiligo or asthma in childhood have been completely relieved, and no intervention in adults can be included; The subjects who needed medical intervention with bronchial dilation were ineligible;
* Patients are using immunity inhibitors or systemic hormone therapy for immunosuppression purpose (such as prednisone > 10 mg/day), except for local hormone therapy.
* Patients were known to be allergic to macromolecular protein, or any components in ipilimumab or SHR-1210;
* Patients with clinical symptoms of central nervous system metastasis (e.g. brain edema, requirement of hormone intervention, or brain metastases progression);
* Another malignancy within 2 years prior to screening, with the exception of adequately treated in-situ carcinoma of the cervix, uteri, basal or squamous cell carcinoma or non-melanomatous skin cancer;
* Patients with congenital or acquired immunodeficiency (such as HIV infection), or active hepatitis (HBV DNA≥10⁴/ml);
* Any severe and / or uncontrolled medical conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-05-15 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety in the treatment of ipilimumab followed by SHR1210 | 24 months
  Adverse events occurring up to 30 days after the last dose of ipilimumab or SHR1210 are evaluated and graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.0.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to 4 weeks
  ORR as measured in accordance with the Response Evaluation Criteria In Solid Tumours (RECIST) version 1.1
Clinical Benefit Response (CBR) | Up to 4 weeks
  CBR as measured in accordance with the Response Evaluation Criteria In Solid Tumours (RECIST) version 1.1
Progression-free Survival (PFS) | Up to 4 weeks
  PFS as measured in accordance with the Response Evaluation Criteria In Solid Tumours (RECIST) version 1.1
Overall survival (OS) | Up to 4 weeks
  OS as measured in accordance with the Response Evaluation Criteria In Solid Tumours (RECIST) version 1.1
Duration of response (DOR) | Up to 4 weeks
  DOR as measured in accordance with the Response Evaluation Criteria In Solid Tumours (RECIST) version 1.1
Time To Progression (TTP) | Up to 4 weeks
  TTP as measured in accordance with the Response Evaluation Criteria In Solid Tumours (RECIST) version 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Cancer Center of Sun-Yat Sen University (CCSYSU), Guangzhou, Guangdong, China